CLINICAL TRIAL: NCT05972096
Title: Clinical Trial of Skills Training for Long Lasting Symptoms in Borderline Personality Disorder
Brief Title: DBT Skills Expanded With Contextual Intervention for Long Lasting Symptoms in Borderline Personality Disorder
Acronym: DBT+Context
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-TLP-2020-104
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Borderline Personality Disorders; BPD
Keywords: borderline personality disorder; long-lasting symptoms; dialectical behavior therapy skills; contextual approach.
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial aims to test the efficacy of this expanded skills DBT-based intervention with self-compassion and contextual-based skills targeting long-lasting BPD compared with treatment as usual.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of DBT-ST, self-compassion, and contextual-based skills. (Experimental): Combination of DBT-ST, self-compassion, and contextual-based skills.
  Interventions: Behavioral: Combination DBT, self-compassion and contextual-based skills
- Control Group (Placebo Comparator): Treatment as usual. Although these individuals did not receive any new specific psychotherapeutic intervention for BPD, they valued the higher frequency of psychiatric visits, attention in crisis, family care, and greater experience and sensitivity in the management of BPD.
  Interventions: Behavioral: Combination DBT, self-compassion and contextual-based skills

INTERVENTIONS:
Behavioral: Combination DBT, self-compassion and contextual-based skills — Psychotherapy combination. Skills of DBT plus self-compassion and contextual skills

SUMMARY:
Although borderline personality disorder (BPD) tend to the clinical remission in long-term follow-up studies, a significant subgroup of patients continues to present long lasting symptoms such as low mood, emptiness and persistent impairment in psychosocial adjustment. The prevalence of this subsample of individuals is considerably increasing last years. New interventions addressed to these individuals are need, the aim of this study is to evaluate the efficacy of a novel intervention combining dialectical behavioral therapy skills training with self-compassion and contextual-based skills for patients with long-lasting BPD.

DETAILED DESCRIPTION:
Sixty individuals with BPD and long lasting symptoms that have been received previously dialectical-behavioral therapy skills training (DBT-ST) will be included in a randomized clinical trial. They will be randomly assigned to receive an add-on skills training intervention involving the combination of DBT-ST, self-compassion, and contextual-based skills for long lasting symptoms versus treatment as usual during 12-weeks. Patients will be evaluated pre and post intervention and 3-month follow-up. The outcome measures are well-being indicators and clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years of age
* Primary diagnosis of BPD according to Diagnostic Statistical Manual IV criteria and by the structured interviews: Diagnosis Structured clinical interview for axis II personality disorders (SCID II; First et al. 1997) and Diagnostic Interview for Borderlines Revised (DIB-R)
* Previous participation in DBT-ST intervention
* Signed informed consent.

Exclusion Criteria:

* Presence of life-threatening behaviors in the last 12 months
* PTSD or related symptoms
* Diagnosis of drug-induced psychosis, organic brain syndrome, bipolar or psychotic disorder
* Intellectual disability
* Participation in any other psychotherapy treatment during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Pemberton Happiness Index (PHI) | 1 month
  Happiness index (minimum 0- maximum 110) Higher scores better

SECONDARY OUTCOMES:
Borderline Symptoms List-23 (BSL-23) | 1 week
  Symptoms of Borderline (minimum 0- maximum 92). Higher scores worse
Remission from Depression Questionnaire (RDQ) | 1 week
  Depression (minimum 0- maximum 84). Higher scores worse
Self Compassion Scale Short Form (SCS-SF) | 1 month
  Compassion scale (12 items, minimum 12- maximum 60). Higher scores worse
Forms of Self-Criticism/Self-Attacking and Self-Reassuring Scale (FSCRS) | 1 month
  Self-criticism forms (14 items, minimum 0- maximum 56). Higher scores worse
Satisfaction with life scale (SWLS) | 1 month
  Well being (5 items, minimum 5 - maximum 25). Higher scores better
Quality of life scale (WHO-QOL_BREF) | 2 weeks
  Quality of life OMS (26 items, minimum 26- maximum 130). Higher scores better

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Soler, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Juan Carlos Pascual Mateos, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No